CLINICAL TRIAL: NCT00282906
Title: [F-18]-Fluorodeoxyglucose (FDG) Positron Emission Tomography and Computed Tomography (PET-CT) in Metastatic Prostate Cancer
Brief Title: FDG Positron Emission Tomography and Computed Tomography (PET-CT) in Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4P-05-1
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-CT (Experimental)
  Interventions: Device: hybrid PET-CT imaging system

INTERVENTIONS:
Device: hybrid PET-CT imaging system — 15 mCi of FDG

SUMMARY:
This is an National Institute of Health (NIH) funded, investigator-initiated, single center prospective study to investigate the ability of the new dual-modality positron emission tomography and computed tomography (PET-CT) imaging systems in comparison to conventional imaging methods in assessing treatment response in men with metastatic prostate cancer. The investigators will enroll two groups of men with stage IV metastatic prostate cancer, each group will be comprised of 160 patients.

* Group I: men with newly diagnosed hormone-responsive measurable metastatic disease who will be treated with androgen-ablation therapy
* Group II: men with newly-developed hormone-refractory measurable metastatic disease who will be treated with chemotherapy and /or other therapies for hormone refractory disease

To be eligible, men in either group must have rising serum prostate specific antigen (PSA) level - defined as at least 2 consecutive rises in PSA documented over a reference value (1st measure within 28 days prior to recruitment). The first rising PSA (2nd measure) should be taken at least 14 days after the reference value. A confirmatory PSA measure (3rd measure) obtained at least 14 days after the 2nd measure is required and must be greater than the 2nd measure. Additionally, patients must have a serum PSA concentration of at least 2 ng/mL in addition to increasing PSA to be eligible. Patients will be followed with the PET-CT at 4, 8, and 12 months after the initiation of androgen ablation therapy (Group I) or chemotherapy (Group II).

DETAILED DESCRIPTION:
Our long-range objective is to obtain pilot data to investigate the ability of the new dual-modality positron emission tomography and computed tomography (PET-CT) imaging systems for assessing treatment response in patients with metastatic prostate cancer in comparison to conventional imaging. PET-CT is not employed here for staging; all men in this study will have stage IV metastatic prostate cancer. We believe that the combined anatomic and in-vivo metabolic imaging information provided by PET-CT allows accurate objective assessment of such critical clinical issues as early prediction and evaluation of response or resistance to various therapeutic interventions, including the novel chemotherapy regimen, as well as the prediction of key clinical outcomes such as time to hormone-refractoriness and survival. Our intermediate-range objective is therefore to investigate the diagnostic and prognostic utility of PET-CT with the most commonly available PET tracer, [F-18]-fluorodeoxyglucose (FDG), in metastatic prostate cancer. We plan to correlate the treatment-induced changes of glucose metabolism in metastatic prostate cancer lesions to the changes in various conventional clinical, laboratory, and diagnostic imaging parameters such as serum prostate-specific antigen level, lesion size, time to androgen independence, and survival. This objective is motivated by our preliminary basic science and clinical data as well as the published reports of other investigators demonstrating the pragmatic potential diagnostic and prognostic utility of FDG PET-CT in men with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Group-I (hormone-responsive) inclusion criteria:

* Age > 21 years, men of all ethnic backgrounds
* Patient must have had a histological diagnosis of adenocarcinoma of prostate and currently must have metastatic disease (stage TxNxM1) that is hormone- naïve received prior to the development of objective evidence for MACRO metastatic or recurrent disease (e.g. during biochemical PSA relapse without imaging evidence of disease).
* Evidence of metastatic disease must be documented as: conventional imaging evidence for metastatic disease as determined by CT, bone scintigraphy, or both (Note: although there are no strict windows for obtaining other scans bone, CT) relative to the timing of the PET scans, every effort will be made to have these 'standard' scans obtained within 3 months of the Baseline PET scan

Group-II (hormone-refractory) inclusion criteria:

* Age > 21 years, men of all ethnic backgrounds
* Patients must have received prior hormonal therapy. Patients treated with orchiectomy are eligible.
* Patient must have had a histological diagnosis of adenocarcinoma of prostate and currently must have metastatic disease (stage TxNxM1) that is unresponsive or refractory to hormonal therapy. Evidence of unresponsive or refractory disease must be documented by either:

  1. a progression of disease assessed with CT or bone scan or as judged clinically based on factors such as increasing bone pain (Note: although there are no strict windows for obtaining other scans (bone, CT) relative to the timing of the PET scans, every effort will be made to have these 'standard' scans obtained within 3 months of the PET scan) OR
  2. a rising serum PSA level - defined as at least 2 consecutive rises in PSA documented over a reference value (1st measure within 3 months prior to recruitment); The first rising PSA (2nd measure) should be taken at least 14 days after the reference value. A confirmatory PSA measure (3rd measure) should be obtained at least 14 days after the 2nd measure and must be greater than the 2nd measure. Additionally, patient must have a serum PSA concentration of at least 2 ng/mL in addition to increasing PSA to be eligible. However, if the patient is clinically judged to have progressive disease irrespective of PSA (e.g. metastasis-related bone pain, clear increase in lesions evident on a bone scan and/or CT if available), documenting a minimum or rising PSA level would not be required.

Other general inclusion criteria for both groups:

* If the treating physician has determined that the patient is not clinically responding to the current therapy prescribed and, in the best interest of the patient, the physician plans to change the treatment to a new treatment.

  1. Example: a Group I patient currently treated with a form of anti-androgen therapy which is not responding; the patient can be considered for enrollment into the PET-CT imaging study prior to a new anti-androgen therapy even though he was treated with anti-androgen therapy before. The wait time between the end of old therapy and the beginning of the new therapy is based entirely on clinical judgment
  2. Example: a Group II patient currently treated with a form of therapy for hormone refractory disease (chemo) therapy which is not responding; the patient can be considered for enrollment into the PET-CT imaging study prior to a new therapy even though he was treated with chemotherapy another type of hormone-refractive therapy before. The wait time between the end of old therapy and the beginning of the new therapy is based entirely on clinical judgment
* May have received prior surgery (14 days must have elapsed since completion of surgery with recovery from side effects)
* Creatinine ≤ 2.5 x the institutional upper limit of normal (within 28 days prior to enrollment)
* Men of childbearing potential must be willing to consent to use effective contraception.
* Must be competent to consent to study requirements
* Patients may also be enrolled in the study from either group if the therapeutic regimen (hormone therapy or chemotherapy and/or other therapies for hormone refractory disease has been administered for up to 2 weeks prior to the baseline PET scan.
* OPTIONAL: Completed analgesic pain survey. If unable to complete questionnaires in English or Spanish, patient can still participate in this study.

Exclusion Criteria:

* History of cancer other than prostate cancer (except squamous cell carcinoma of the skin that has been treated with curative intent) or other cancers clinically judged to be cured or inactive based on history, physical examination, tumor markers, or imaging findings.
* Active infection (except mild upper respiratory infections or other sites if clinically judged not to interfere with image interpretation on a per case basis)
* History of poorly-controlled diabetes mellitus (with Fasting Blood Glucose greater than 200 mg/dL) - in order to avoid false negative results due to glucose competition with [F-18]-Fluorodeoxyglucose in cellular uptake
* Active inflammatory conditions (e.g. rheumatoid arthritis, sarcoid)
* History of complicated non-healing fracture
* Not competent to consent

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2005-10-03 (Actual); Primary Completion 2013-12-19 (Actual); Study Completion 2014-08-19 (Actual)

PRIMARY OUTCOMES:
PET/CT imaging validity | every 4 months

SECONDARY OUTCOMES:
Response | every 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Jadvar, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Jadvar H, Desai B, Ji L, Conti PS, Dorff TB, Groshen SG, Pinski JK, Quinn DI. Baseline 18F-FDG PET/CT parameters as imaging biomarkers of overall survival in castrate-resistant metastatic prostate cancer. J Nucl Med. 2013 Aug;54(8):1195-201. doi: 10.2967/jnumed.112.114116. Epub 2013 Jun 19. PMID 23785174